CLINICAL TRIAL: NCT06430060
Title: The Clinical Investigation of Colgate Dual Zinc Toothpaste as Compared to Colgate Cavity Protection Toothpaste in Controlling Established Plaque and Gingivitis (A Threemonth Clinical Study)
Brief Title: The Clinical Investigation of Colgate Dual Zinc Toothpaste as Compared to Colgate Cavity Protection Toothpaste in Controlling Established Plaque and Gingivitis
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRO-2024-03-GIN-DZN-CN-YPZ
Record Dates: First submitted 2024-05-21; First posted 2024-05-28 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Plaque, Dental; Gingivitis
MeSH Terms: conditions — Dental Plaque; Gingivitis | interventions — green tea bioflavonoid, zinc ascorbate-containing toothpaste

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Colgate Dual Zinc Toothpaste (Experimental): toothpaste
  Interventions: Drug: zinc containing toothpaste
- Colgate Cavity Protection Toothpaste (Active Comparator): toothpaste
  Interventions: Drug: MFP Fluoride toothpaste

INTERVENTIONS:
Drug: zinc containing toothpaste — Toothpaste
  Arms: Colgate Dual Zinc Toothpaste
Drug: MFP Fluoride toothpaste — toothpaste
  Arms: Colgate Cavity Protection Toothpaste

SUMMARY:
Qualified subjects will be enrolled and randomized to either one of the two study groups described above based on their initial Plaque and Gingivitis scores. Subjects will be instructed to use the products according to the instructions provided. Subjects will return to the dental office for evaluation after three months of product use. All subjects will be followed for adverse events throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects, ages 18-70, inclusive.
* Availability for the three-month duration of the clinical research study.
* Good general health.
* Minimum of 20 uncrowned permanent natural teeth (excluding third molars).
* Initial gingivitis index of at least 1.0 as determined by the use of the Loe and Silness Gingival Index.
* Initial plaque index of at least 1.5 as determined by the use of the Quigley and Hein Plaque Index (Turesky Modification).
* Signed Informed Consent Form

Exclusion Criteria:

* Presence of orthodontic bands.
* Presence of partial removable dentures.
* Tumor(s) of the soft or hard tissues of the oral cavity.
* Advanced periodontal disease (purulent exudate, tooth mobility, and/or extensive loss of periodontal attachment or alveolar bone).
* Five or more carious lesions requiring immediate restorative treatment.
* Antibiotic use any time during the one month prior to entry into the study.
* Participation in any other clinical study or test panel within the one month prior to entry into the study.
* Dental prophylaxis during the past two weeks prior to baseline examinations.
* History of allergies to oral care/personal care consumer products or their ingredients.
* On any prescription medicines that might interfere with the study outcome.
* An existing medical condition which prohibits eating or drinking for periods up to 4 hours.
* History of alcohol or drug abuse.
* Pregnant or lactating subjects

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Loe-Silness Gingival Index score | baseline, 2 week, 6 week, 3 month
  A Loe-Silness Gingival Index score from 0 to 3 will be assigned by the examining dentist to all scoreable surfaces of the maxillary and mandibular teeth using a dental light and dental mirror. A whole mouth mean score for each subject will be determined by adding the values given by the examining dentist to each scoreable surface and dividing that number by the total number of surfaces scored.
Quigley-Hein Plaque Index score | baseline, 2 week, 6 week, 3 month
  A Quigley-Hein Plaque Index score of 0 to 5 will be assigned to all scoreable disclosed surfaces of the maxillary and mandibular teeth using a dental light and dental mirror. A whole mouth score for each subject will be determined by adding the values given by the dental examiner to each scoreable surface and dividing that number by the total number of surfaces scored.

CONTACTS AND LOCATIONS:
Overall Officials: Deyu Hu, DDS, MS, Principal Investigator — West China Dental Institute of Chengdu
Locations (1):
- West China Dental Institute of Chengdu, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No